CLINICAL TRIAL: NCT01197924
Title: Médulloblastome of the Child and After-effects Cognitive: Study Anatomo-functional by IRM of the Working Memory
Brief Title: MEDIR Medulloblastome
Acronym: MEDIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: PAGNIER Anne, Professor, Pédiatrie
Other Study IDs: 07PHN01
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Child Cancer Brain
Keywords: child cancer brain

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy volonteer children: paired for the sex and the age
  Interventions: Other: IRMf Bold
- older children followed for a médulloblastome cérébelleux: children followed for a médulloblastome treaty by surgery, radiotherapy and chemotherapy
  Interventions: Other: IRMf Bold

INTERVENTIONS:
Other: IRMf Bold — IRMf BOLD of the working memory

SUMMARY:
The medulloblastome is a tumour of the child relatively frequent usually sitting in the cerebellum and treated by surgery, radiotherapy and chemotherapy. After the treatment, these children present cognitive disorders and in particular disorders of the working memory associated with a fall with the school performances. By studying a troop of 32 children, we could show that the disorders of the working memory prevail during the handling of information presented visually and with verbal contents. However, the specific engagement of the cerebellum in the tasks of working memory according to the sensory method of presentation (visual or auditive) and the nature (verbal or not verbal) of information to treat vague remainder. Moreover, the anatomical attacks associated with these disorders remain ignored in these children. The best comprehension of the bases anatomo-functional calculuses which underlie their cognitive deficits is essential to develop new strategies of treatment and rehabilitation.

Objectives:

* To describe in IRMf of the common and specific networks engaged during the execution of the tasks of working memory according to the sensory type and the nature of information to be memorized.
* To describe in IRMf the cortical reorganizations necessary to the execution of the mnemic tasks among patients.
* To describe in anatomical IRM and of the tensor of diffusion lesions cérébelleuses and cerebral, cortical and subcortical associated with these disorders.
* To study the correlations radio-private clinics between data IRM and the data neurological and neuropsychological of the children explored according to protocol ONCORAP

DETAILED DESCRIPTION:
The functional study should make it possible to show the specifically committed networks according to the cognitive tasks. Among patients, the relative difficulty to carry out the tasks of working memory should be accompanied by a recruitment of the dorso-side cortex préfrontal, lower and parietal frontal cortex but also of the median frontal areas such as the additional driving surface, the former cingulum. Moreover, one deterioration of the engagement of the cérébello-cerebral network (left lower parietal cortex and cérébelleux cortex lower right) facilitating the execution of these tasks should be observed.

ELIGIBILITY:
Inclusion Criteria:

* Old from 8 to 12 years
* Total IQ > 70 for the participation in the study and/or age développemental 7 years minimum
* Treaties for a médulloblastome after the 6 years age in remission supplements with 6 months a minimum time compared to the end of all the treatments
* Followed within the framework of the protocol of evaluation of the mnemic and attentionnelles after-effects
* Sensory after-effects compatible with the realization of the tasks and good performances at the time of the preceding drive the IRM
* Absence of counter-indication to the IRM
* Absence of catch of méthylphénidate (Ritaline®) for the treatment of disorders attentionnels 48h before the IRM
* Enlightened assent signed by at least one of the two parents or holders of the parental authority and by the child (minor)

Exclusion Criteria:

* Agitation or movements of the head at the time the IRM
* Artifacts of magnetic susceptibility in projection of the areas of interest (intracranial haemorrhage, cortical and/or metal remains post-operative) • Bad execution of the cognitive tasks
* Tumoral relapse in the course of protocol

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: child Treaties for a médulloblastome after the 6 years age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anne A PAGNIER, Doctor, Principal Investigator — University Hospital, Grenoble
Locations (8):
- France (8):
  - University hospital, Bordeaux, Bordeaux
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon, Lyon
  - Hôpital Frédéric Joliot Orsay - Hôpital Necker, Paris, Paris
  - Institut Curie, Paris, Paris
  - University Hospital, Saint-Etienne, Saint Etienne
  - Institut Gutave Roussy, Villejuif, Villejuif
  - SMAEC, Villeurbanne, Villeurbanne
  - UniversityHospitalGrenoble, Grenoble